CLINICAL TRIAL: NCT03419858
Title: The Role of Endogenous Opioidergic Systems in Breathing Based Analgesia
Brief Title: The Role of Opioidergic Systems in Breathing Based Analgesia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Fadel Zeidan, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00040519
Record Dates: First submitted 2018-01-16; First posted 2018-02-05 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Pain
Keywords: Pain; Slow-Breathing; Mindfulness; Opioids; Placebo
MeSH Terms: conditions — Pain; Hypoventilation | interventions — Mindfulness; Naloxone; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The study employed a double blind 3x2x2 crossover factorial design. Baseline pain intensity and pain unpleasantness ratings were assessed using visual analog scales (11 point) obtained before and after four, 5-minute noxious heat stimulation series (49°C). Study volunteers (20/group; 60 total) were randomized and subsequently participated in a four session (20min/session) mindfulness meditation, placebo-meditation, or slow-breathing training regimen. After training completion, subjects reported to the Wake Forest Clinical Research Unit to test the study hypotheses across two separate experimental sessions. Half of the study volunteers (n=10) from each group were administered naloxone (opioid antagonist; 0.15 mg/kg bolus+ 0.1mg/kg/hour infusion) and in the subsequent session were administered IV placebo-saline and vice versa.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the study physician, research coordinator, and research pharmacist were aware of drug assignments. Research staff (nurses; research technicians) and the PI were not blinded to drug assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Mindfulness Meditation Group (Experimental): Subjects participated in four sessions (20 min/session) of mindfulness training. Participants were taught that perceived sensory events are "momentary" and "fleeting" and require no further evaluation. They were asked to close their eyes, relax and to focus on the flow of their breathing and "simply let go" of discursive thoughts.
  Interventions: Behavioral: Mindfulness Meditation; Drug: Naloxone; Other: Saline
- Placebo Meditation Group (Active Comparator): The purpose of this intervention was to lead subjects to attend to one's breathing in a non-evaluative manner. Subjects were instructed to sit with a straight posture, closed eyes, and to take a deep, slow breaths every 2-3 minutes.
  Interventions: Behavioral: Placebo Meditation; Drug: Naloxone; Other: Saline
- Slow-Breathing Group (Active Comparator): A validated (Chalaye et al., 2009) slow breathing training regimen was employed, using fluctuating light, to teach individuals to independently lower their respective respiration rate. Subjects practiced lowering their respiration rates across four, 20 minute sessions.
  Interventions: Behavioral: Slow-Breathing; Drug: Naloxone; Other: Saline

INTERVENTIONS:
Behavioral: Mindfulness Meditation — A well-validated brief mindfulness-based mental training regimen [four sessions; 20 min/session] was used to teach patients to independently practice mindfulness meditation.
  Other Names: mental training
  Arms: Mindfulness Meditation Group
Behavioral: Placebo Meditation — A well-validated brief meditation-based mental training regimen [four sessions; 20 min/session] was used to teach patients to independently practice closing their eyes and take a deep breath every few minutes.
  Other Names: mental training
  Arms: Placebo Meditation Group
Behavioral: Slow-Breathing — Study volunteers practiced lowering their breathing rate, across four, 20 minute training sessions, in response to a fluctuating light with the guidance of a trained facilitator.
  Other Names: mental training
  Arms: Slow-Breathing Group
Drug: Naloxone — A 0.15 mg/kg bolus dose of naloxone (Naloxone Hydrichloride, Amphastar Pharmaceuticals, Inc., Rancho Cucamonga, California) in 25ml normal saline was administered over 10 minutes. We also administered a supplementary IV infusion dose of 0.1mg/kg/hour naloxone immediately after bolus infusion ceased till the end of the experiment.
Other: Saline — A 0.15 mg/kg bolus dose of saline in 25ml normal saline was administered over 10 minutes. We also administered a supplementary IV infusion dose of 0.1mg/kg/hour saline immediately after bolus infusion ceased till the end of the experiment.

SUMMARY:
The purpose of this psychophysical and pharmacologic study is to determine if slow-breathing induced pain relief is mediated by endogenous opioids in response to intravenous (IV) administration of the opioid antagonist naloxone during noxious heat stimulation. We were also interested in disentangling the endogenous analgesic mechanisms supporting mindfulness-based analgesia.

DETAILED DESCRIPTION:
The proposed study will employ a graded analytical approach to compare mindfulness to placebo-meditation and a slow-breathing exercise in response to double-blind intravenous administration (IV) of naloxone/placebo-saline and noxious heat stimulation. The aim of this study is to determine if slow-breathing induced analgesia is associated with the release of endogenous opioids. The proposed study will disentangle the specific stage of cognitive and/or respiration-based involvement (if any) of opioidergically mediated pain relief, a critical step in identifying the specific analgesic mechanisms corresponding to mindfulness based cognitive techniques.

ELIGIBILITY:
Inclusion Criteria:

* Normal volunteers with no history of chronic pain problems
* Volunteers had no prior meditation experience
* Volunteers could be male and non-pregnant females.
* Volunteers of all ethnic backgrounds were included.

Exclusion Criteria:

* Female volunteers could not be pregnant.
* They could not be taking opioids or antidepressants.
* Subjects with a repeated history of syncope, loss of consciousness, light headedness, nausea, dizziness, or vomiting in response to needles or blood could not participate in the study.
* Subject could not be using exogenous opiates for the complete duration of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2017-06-27 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale Pain intensity and Unpleasantness ratings as a function of each respective cognitive manipulations and activation in response to naloxone and/or saline. | Up to 3 weeks
  The visual analog scale (VAS) measures pain ratings that are assessed in response to noxious (49°C) thermal stimuli applied to the back of the right calf muscle.
  Pain intensity and unpleasantness ratings will be assessed with a Visual Analog Scale. The minimum rating ("0") is designated as "no pain" whereas the maximum ("10") is labeled as "most intense imaginable" or "most unpleasant imaginable". Higher values corresponded to higher perceived pain ratings.
  Pain ratings were assessed at baseline (session 1) and again at sessions six and seven to determine the impact of the mental training regimens. At session six and seven, subjects were given an infusion of either naloxone or saline to address the potential contribution of the opioidergic system in the cognitive modulation of pain.

SECONDARY OUTCOMES:
Respiration Rate Measures | Up to 3 weeks
  A respiratory transducer (TSD 201; Biopac Systems) was placed around the chest to measure the participant's rate of respiration.
State Anxiety Inventory | up to 3 weeks
  This inventory is a 20 question test used to measure a subject's state of anxiety. A numeric value between 1 (Not at all) and 4 (Very Much So) is provided in response to each statement. The range of scores for this test is between 20 and 80, with higher scores reflecting higher estimates of anxiety.
Pain Catastrophizing Scale (PCS) | up to 3 weeks
  The PCS is a 13 item scale, with each item rated on a 5-point scale between: 0 (Not at all) and 4 (all the time). The PCS is broken into three subscales including: magnification, rumination, and helplessness. The total range of scores is between 0-52 with higher values reflecting more salient impacts of pain on one's day to day experience.
Cohen Perceived Stress Scale (CPS) | up to 3 weeks
  The CPS is a series of 10 temporally constrained (i.e. in the last month) questions meant to ascertain the relative frequency of stressors in one's life, ranging from never (scored as 0) to very often (scored as 4). All positively stated questions are reversed scored and then all items are summed to yield a final estimate of stress. The higher the score the higher the level of stress.
Treatment Effectiveness Scale | up to 3 weeks
  A VAS assessed the effectiveness of the study's intervention. Values on this scale vary continuously between 0 (not effective) and 10 (most effective imaginable). Higher values indicate a subject's greater confidence in the perceived treatment effectiveness.
Attitude Toward Treatment Scale (ATTS) | up to 3 weeks
  The ATTS was used to monitor a participant's impressions and attitudes about the interventions used in this study. It supplies 5 multiple-choice questions answered on a 10 point scale, ranging from 0 (not logical) to 9 (very logical). Higher scores reflect more positive subject impressions about the therapeutic interventions.
Center for Epidemiological Studies Depression Scale (CES-D) | up to 3 weeks
  This is a brief self-report questionnaire used to measure the severity of depressive symptoms. The CES-D is an inventory of 20 self-report items regarding depressive symptoms. Each question is graded on a 0 to 3 point scale with 0 representing "not at all" and 3 representing "a lot". Four questions (4,8,12, and 16) are reverse scored. A score of 15 or higher indicates a risk for depression.
Stress-Level Visual Analogue Scale | up to 3 weeks
  A VAS was employed to measure subjective stress ratings. Values on this scale vary continuously between 0 (no stress) to 10 (most stress imaginable). Higher values indicate higher assessments of the subject's stress level.
Naloxone Symptom Assessments | Up to 3 weeks
  A numerical ratings scale was used to assess potential naloxone related symptomology after each clinical research unit session. "0" was designated as "non-existent" and "6" was characterized as "extremely strong". We measured symptoms corresponding to "dry mouth, dry skin, blurred vision, sedation, nausea, dizziness, and headache."

CONTACTS AND LOCATIONS:
Overall Officials: Fadel Zeidan, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Apkarian AV, Bushnell MC, Treede RD, Zubieta JK. Human brain mechanisms of pain perception and regulation in health and disease. Eur J Pain. 2005 Aug;9(4):463-84. doi: 10.1016/j.ejpain.2004.11.001. Epub 2005 Jan 21. PMID 15979027
- [Background] Bertisch SM, Wee CC, Phillips RS, McCarthy EP. Alternative mind-body therapies used by adults with medical conditions. J Psychosom Res. 2009 Jun;66(6):511-9. doi: 10.1016/j.jpsychores.2008.12.003. Epub 2009 Mar 3. PMID 19446710
- [Background] Borras MC, Becerra L, Ploghaus A, Gostic JM, DaSilva A, Gonzalez RG, Borsook D. fMRI measurement of CNS responses to naloxone infusion and subsequent mild noxious thermal stimuli in healthy volunteers. J Neurophysiol. 2004 Jun;91(6):2723-33. doi: 10.1152/jn.00249.2003. PMID 15136603
- [Background] Brown CA, Jones AKP. Meditation experience predicts less negative appraisal of pain: electrophysiological evidence for the involvement of anticipatory neural responses. Pain. 2010 Sep;150(3):428-438. doi: 10.1016/j.pain.2010.04.017. Epub 2010 May 21. PMID 20494517
- [Background] Chalaye P, Goffaux P, Lafrenaye S, Marchand S. Respiratory effects on experimental heat pain and cardiac activity. Pain Med. 2009 Nov;10(8):1334-40. doi: 10.1111/j.1526-4637.2009.00681.x. Epub 2009 Aug 7. PMID 19671085
- [Background] Clarke TC, Black LI, Stussman BJ, Barnes PM, Nahin RL. Trends in the use of complementary health approaches among adults: United States, 2002-2012. Natl Health Stat Report. 2015 Feb 10;(79):1-16. PMID 25671660
- [Background] Coghill RC, McHaffie JG, Yen YF. Neural correlates of interindividual differences in the subjective experience of pain. Proc Natl Acad Sci U S A. 2003 Jul 8;100(14):8538-42. doi: 10.1073/pnas.1430684100. Epub 2003 Jun 24. PMID 12824463
- [Background] Cusens B, Duggan GB, Thorne K, Burch V. Evaluation of the breathworks mindfulness-based pain management programme: effects on well-being and multiple measures of mindfulness. Clin Psychol Psychother. 2010 Jan-Feb;17(1):63-78. doi: 10.1002/cpp.653. PMID 19911432
- [Background] Eippert F, Bingel U, Schoell ED, Yacubian J, Klinger R, Lorenz J, Buchel C. Activation of the opioidergic descending pain control system underlies placebo analgesia. Neuron. 2009 Aug 27;63(4):533-43. doi: 10.1016/j.neuron.2009.07.014. PMID 19709634
- [Background] Friesner SA, Curry DM, Moddeman GR. Comparison of two pain-management strategies during chest tube removal: relaxation exercise with opioids and opioids alone. Heart Lung. 2006 Jul-Aug;35(4):269-76. doi: 10.1016/j.hrtlng.2005.10.005. PMID 16863899
- [Background] Grant JA, Rainville P. Pain sensitivity and analgesic effects of mindful states in Zen meditators: a cross-sectional study. Psychosom Med. 2009 Jan;71(1):106-14. doi: 10.1097/PSY.0b013e31818f52ee. Epub 2008 Dec 10. PMID 19073756
- [Background] Grant JA, Courtemanche J, Duerden EG, Duncan GH, Rainville P. Cortical thickness and pain sensitivity in zen meditators. Emotion. 2010 Feb;10(1):43-53. doi: 10.1037/a0018334. PMID 20141301
- [Background] Grill JD, Coghill RC. Transient analgesia evoked by noxious stimulus offset. J Neurophysiol. 2002 Apr;87(4):2205-8. doi: 10.1152/jn.00730.2001. PMID 11929939
- [Background] Kabat-Zinn J. An outpatient program in behavioral medicine for chronic pain patients based on the practice of mindfulness meditation: theoretical considerations and preliminary results. Gen Hosp Psychiatry. 1982 Apr;4(1):33-47. doi: 10.1016/0163-8343(82)90026-3. PMID 7042457
- [Background] Kabat-Zinn J, Lipworth L, Burney R. The clinical use of mindfulness meditation for the self-regulation of chronic pain. J Behav Med. 1985 Jun;8(2):163-90. doi: 10.1007/BF00845519. PMID 3897551
- [Background] Koyama T, McHaffie JG, Laurienti PJ, Coghill RC. The single-epoch fMRI design: validation of a simplified paradigm for the collection of subjective ratings. Neuroimage. 2003 Jul;19(3):976-87. doi: 10.1016/s1053-8119(03)00119-8. PMID 12880826
- [Background] Ludwig DS, Kabat-Zinn J. Mindfulness in medicine. JAMA. 2008 Sep 17;300(11):1350-2. doi: 10.1001/jama.300.11.1350. No abstract available. PMID 18799450
- [Background] Lutz A, Slagter HA, Dunne JD, Davidson RJ. Attention regulation and monitoring in meditation. Trends Cogn Sci. 2008 Apr;12(4):163-9. doi: 10.1016/j.tics.2008.01.005. Epub 2008 Mar 10. PMID 18329323
- [Background] MacLean KA, Ferrer E, Aichele SR, Bridwell DA, Zanesco AP, Jacobs TL, King BG, Rosenberg EL, Sahdra BK, Shaver PR, Wallace BA, Mangun GR, Saron CD. Intensive meditation training improves perceptual discrimination and sustained attention. Psychol Sci. 2010 Jun;21(6):829-39. doi: 10.1177/0956797610371339. Epub 2010 May 11. PMID 20483826
- [Background] Martin SL, Kerr KL, Bartley EJ, Kuhn BL, Palit S, Terry EL, DelVentura JL, Rhudy JL. Respiration-induced hypoalgesia: exploration of potential mechanisms. J Pain. 2012 Aug;13(8):755-63. doi: 10.1016/j.jpain.2012.05.001. Epub 2012 Jul 4. PMID 22770894
- [Background] Martucci KT, Eisenach JC, Tong C, Coghill RC. Opioid-independent mechanisms supporting offset analgesia and temporal sharpening of nociceptive information. Pain. 2012 Jun;153(6):1232-1243. doi: 10.1016/j.pain.2012.02.035. Epub 2012 Apr 13. PMID 22503222
- [Background] Mehling WE, Hamel KA, Acree M, Byl N, Hecht FM. Randomized, controlled trial of breath therapy for patients with chronic low-back pain. Altern Ther Health Med. 2005 Jul-Aug;11(4):44-52. PMID 16053121
- [Background] Price DD. Psychological and neural mechanisms of the affective dimension of pain. Science. 2000 Jun 9;288(5472):1769-72. doi: 10.1126/science.288.5472.1769. PMID 10846154
- [Background] Price DD, McHaffie JG, Larson MA. Spatial summation of heat-induced pain: influence of stimulus area and spatial separation of stimuli on perceived pain sensation intensity and unpleasantness. J Neurophysiol. 1989 Dec;62(6):1270-9. doi: 10.1152/jn.1989.62.6.1270. PMID 2600624
- [Background] Price DD, Bush FM, Long S, Harkins SW. A comparison of pain measurement characteristics of mechanical visual analogue and simple numerical rating scales. Pain. 1994 Feb;56(2):217-226. doi: 10.1016/0304-3959(94)90097-3. PMID 8008411
- [Background] Rhudy JL. Respiration-induced hypoalgesia: additional evidence for pain modulation deficits in fibromyalgia? Pain. 2010 Apr;149(1):1-2. doi: 10.1016/j.pain.2010.01.004. Epub 2010 Feb 1. No abstract available. PMID 20122804
- [Background] Rosier EM, Iadarola MJ, Coghill RC. Reproducibility of pain measurement and pain perception. Pain. 2002 Jul;98(1-2):205-16. doi: 10.1016/s0304-3959(02)00048-9. PMID 12098633
- [Background] Schoell ED, Bingel U, Eippert F, Yacubian J, Christiansen K, Andresen H, May A, Buechel C. The effect of opioid receptor blockade on the neural processing of thermal stimuli. PLoS One. 2010 Aug 27;5(8):e12344. doi: 10.1371/journal.pone.0012344. PMID 20811582
- [Background] Stone CI, Demchik-Stome DA, Horan JJ. Coping with pain: a component analysis of Lamaze and cognitive-behavioral procedures. J Psychosom Res. 1977;21(6):451-6. doi: 10.1016/0022-3999(77)90067-8. No abstract available. PMID 599507
- [Background] Tracey I, Mantyh PW. The cerebral signature for pain perception and its modulation. Neuron. 2007 Aug 2;55(3):377-91. doi: 10.1016/j.neuron.2007.07.012. PMID 17678852
- [Background] Wells RE, Bertisch SM, Buettner C, Phillips RS, McCarthy EP. Complementary and alternative medicine use among adults with migraines/severe headaches. Headache. 2011 Jul-Aug;51(7):1087-97. doi: 10.1111/j.1526-4610.2011.01917.x. Epub 2011 Jun 7. PMID 21649654
- [Background] Zautra AJ, Fasman R, Davis MC, Craig ADB. The effects of slow breathing on affective responses to pain stimuli: an experimental study. Pain. 2010 Apr;149(1):12-18. doi: 10.1016/j.pain.2009.10.001. Epub 2010 Jan 15. PMID 20079569
- [Background] Zeidan F, Gordon NS, Merchant J, Goolkasian P. The effects of brief mindfulness meditation training on experimentally induced pain. J Pain. 2010 Mar;11(3):199-209. doi: 10.1016/j.jpain.2009.07.015. Epub 2009 Oct 22. PMID 19853530
- [Background] Zeidan F, Johnson SK, Gordon NS, Goolkasian P. Effects of brief and sham mindfulness meditation on mood and cardiovascular variables. J Altern Complement Med. 2010 Aug;16(8):867-73. doi: 10.1089/acm.2009.0321. PMID 20666590
- [Background] Zeidan F, Johnson SK, Diamond BJ, David Z, Goolkasian P. Mindfulness meditation improves cognition: evidence of brief mental training. Conscious Cogn. 2010 Jun;19(2):597-605. doi: 10.1016/j.concog.2010.03.014. Epub 2010 Apr 3. PMID 20363650
- [Background] Zeidan F, Martucci KT, Kraft RA, McHaffie JG, Coghill RC. Neural correlates of mindfulness meditation-related anxiety relief. Soc Cogn Affect Neurosci. 2014 Jun;9(6):751-9. doi: 10.1093/scan/nst041. Epub 2013 Apr 24. PMID 23615765
- [Background] Zeidan F, Martucci KT, Kraft RA, Gordon NS, McHaffie JG, Coghill RC. Brain mechanisms supporting the modulation of pain by mindfulness meditation. J Neurosci. 2011 Apr 6;31(14):5540-8. doi: 10.1523/JNEUROSCI.5791-10.2011. PMID 21471390
- [Background] Zeidan F, Emerson NM, Farris SR, Ray JN, Jung Y, McHaffie JG, Coghill RC. Mindfulness Meditation-Based Pain Relief Employs Different Neural Mechanisms Than Placebo and Sham Mindfulness Meditation-Induced Analgesia. J Neurosci. 2015 Nov 18;35(46):15307-25. doi: 10.1523/JNEUROSCI.2542-15.2015. PMID 26586819
- [Background] Zeidan F, Adler-Neal AL, Wells RE, Stagnaro E, May LM, Eisenach JC, McHaffie JG, Coghill RC. Mindfulness-Meditation-Based Pain Relief Is Not Mediated by Endogenous Opioids. J Neurosci. 2016 Mar 16;36(11):3391-7. doi: 10.1523/JNEUROSCI.4328-15.2016. PMID 26985045
- [Background] Zubieta JK, Bueller JA, Jackson LR, Scott DJ, Xu Y, Koeppe RA, Nichols TE, Stohler CS. Placebo effects mediated by endogenous opioid activity on mu-opioid receptors. J Neurosci. 2005 Aug 24;25(34):7754-62. doi: 10.1523/JNEUROSCI.0439-05.2005. PMID 16120776

DOCUMENTS (1):
  • Statistical Analysis Plan (2016-08-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT03419858/SAP_000.pdf